CLINICAL TRIAL: NCT01231087
Title: Energy Expenditure in Patients Pre and Post Bariatric Surgery
Brief Title: Energy Expenditure Pre and Post Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Gastrocirurgia, Brazil (Other)
Responsible Party: Silvia Leite Faria, Gastrocirurgia
Other Study IDs: Gastrocirurgia
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-10

CONDITIONS: Bariatric Surgery
Keywords: energy expenditure; morbid obesity; bariatric surgery; nutritional follow-up
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Obese patients are going to be submitted to indirect calorimetry pre-operatively and we are going to repeat the same exam 6 months after bariatric surgery (post Roux-en-Y gastric Bypass surgery). They are going to do also body composition analysis in both moments.

The investigators are going to compare the results to see if the bariatric surgery increases their energy expenditure.

ELIGIBILITY:
Inclusion Criteria:

* obese patients that will be submitted to bariatric procedure

Exclusion Criteria:

* patients that don´t have clinical conditions to be submitted to a bariatric procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese petiets
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2008-01; Primary Completion 2008-01 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gastrocirurgia, Brasília, Federal District, Brazil